CLINICAL TRIAL: NCT03869021
Title: Technical Notes on Novel Technique and Step by Step Construction of Computer Guided for Mandibular Distraction Osteogenesis
Brief Title: Computer Guided for Mandibular Distraction Osteogenesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yasser Mohamed Nabil Ahmed Khirat El Hadidi (Other)
Responsible Party: Sponsor-Investigator, Yasser Mohamed Nabil Ahmed Khirat El Hadidi, Assistant Lecturer, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 392B
Record Dates: First submitted 2019-03-01; First posted 2019-03-11 (Actual); Last update posted 2019-03-11 (Actual); Status verified 2019-03

CONDITIONS: Hemifacial Microsomia
Keywords: Computer guided surgery; Hemifacial Microsomia
MeSH Terms: conditions — Goldenhar Syndrome

STUDY DESIGN:
Intervention Model Description: Case control trial
Who Masked: Participant, Care Provider
Masking Description: Single blinding
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Computer guided surgery (Active Comparator): A surgical guide is 3d printed to guide through the surgery, the patients of this group will have the distraction surgery by a guide designed by Mimics 19.0, Materialise NV,Belgium
  Interventions: Other: 3D printed surgical guide constructed
- No surgical guide (free hand surgery) (Other): control group added to investigate the effect of surgical guide
  Interventions: Other: free hand surgery

INTERVENTIONS:
Other: 3D printed surgical guide constructed — A printed surgical guide ( to direct through the surgery and make results predictable), the guide is designed by Mimics 19.0, Materialise NV,Belgium and printed with self cure resin
  Arms: Computer guided surgery
Other: free hand surgery — A control group in which patients are randomly assigned and surgeries are planned without surgical guides and performed free handed
  Arms: No surgical guide (free hand surgery)

SUMMARY:
Objectives: Distraction Osteogenesis is an integral part in management of mandibular defects associated with Hemifacial Microsomia (HFM) and post-ankylotic mandibular defects. The most difficult part in distraction osteogenesis is the prediction of distraction vector and risk of injury to vital structures as inferior alveolar. The current study aimed to present Three-Dimensionally Constructed Computer Guided Splints in Distraction Osteogenesis to get an ideal vector and minimal risk of vital structures injury.

Methods: The study presents computer-guided distraction osteogenesis surgery using prefabricated splints.

DETAILED DESCRIPTION:
The current study was performed on a case control trial of patients complaining of hemifacial microsomia.. The research was reviewed by the ethical committee of the authors institute (approval number: 392, date: 30/12/2015). Written informed consent for the case to be published (incl. images, case history and data) was obtained from the patients for publication of this case report, including accompanying images In order to accurately analyse the patients' condition and formulate an optimal treatment plan, a pre-operative CBCT scan was performed using i-CAT CBCT scanner (Imaging Sciences International, Hatfield, PA, U.S.A).

Each patient was positioned in the machine and imaged at the same manner according to the recommendations of CBCT manufacturer. The Frankfurt plane was positioned parallel to the horizontal plane and the midsagittal plane was perpendicular to the horizontal plane.

The CBCT scan was required to fulfill the following criteria:

* Showing the full bony facial structures, extending from at least the inferior border of the mandible to the supraorbital ridge.
* CBCT scan should be free from any motion artifacts.
* Patient biting on cotton rolls in order to free the occlusion.
* A scan of optimum quality and resolution. (0.25 mm voxel size) IV. Virtual Treatment Planning
* The data from the CBCT scan were exported from the i-CAT Vision software in DICOM format, which was in turn imported into Mimics Medical 19.0 software (Materialise NV, Technologielaan 15, 3001 Leuven, Belgium) for virtual treatment planning.
* Using the "Thresholding" tool, the range of gray value sets is chosen to highlight the mineralized structures and separate them from the rest of soft tissue structures in the scan creating a new mask.
* Using the "Calculate 3D" tool on the new mask, a 3D rendering of the facial mineralized structures is created and is then refined using the "Smoothing" and "Wrap" tools.
* In order to properly orient the patient's head position, analyze the deficiencies, and standardize the planning process, the Frankfort Horizontal plane and the Midsagittal plan were constructed. Frankfort Horizontal Plane was defined by marking the right and left Orbitale, and the Porion of the non-affected side. The Midsagittal plane was defined by marking the Sella, the Nasion, and the Anterior Nasal Spine.
* Using the "Multiple Slice Edit" and "Region Growing" tools when needed, the jaws are separated and the mandible and maxilla are segmented separately.
* Using the "Distraction Wizard", an appropriate distraction type is selected. A distractor is selected and placed on the proposed site for distraction. The osteotomy and vector are visualized and the distractor is activated. This process is repeated until the final outcome is satisfactory. The ideal final outcome is when the canted occlusal plane is corrected and the mandibular midline is coincident with the facial midline simultaneously.
* Using the "Cylinder" tool in the "Medcad" menu, virtual distractor pins and osteotomy disk are drawn to match our selected custom-made distractor. The number of pins, their size, and orientation differed according to the vital structures in each distraction site. Hence, custom-made distractors were used. Guide fixation screws are also added to provide further retention for the guide when needed. The fixation screws, osteotomy and distractor pins are placed so as to avoid injury to any vital structures as the Inferior Alveolar Nerve, tooth buds, and dental roots .
* Using different Boolean operation, the body of the final guide is designed to fit over the bones and teeth and incorporate the different distractor components. It is then exported into STL format.
* The exported STL file is printed with Formlabs Form 2 stereolithography (SLA) 3D printer (Formlabs Inc. Somerville, MA 02143 USA) using Clear Photopolymer resin (FLGPCL02). The finished printed model is then checked for fit with the distractor.
* Prior to surgery, the guide is submerged in a basin containing 2.4% activated glutaraldehyde solution (Cidex) for 20 minutes for high level disinfection.

Surgical Procedure

* The patient was placed in supine position. General anesthesia was administered through Naso-Tracheal intubation. A cannula was inserted in a peripheral vein (18G) and normal saline infusion was started at a rate of 6 ml/kg along with Ringer's solution.
* Anesthesia was induced with IV propofol 1.5-2 mg/kg, fentanyl 1.3 μ/kg and succinyl choline 1mg/kg to facilitate nasotracheal intubation using armored tube. Anesthesia was maintained with isoflurane in oxygen and atracurium in a dose of 0.3-0.6 mg/kg.
* The surgical sites were prepared with povidone iodine and then draped according to the standard oral and maxillofacial surgery operating room procedures.
* An Antibiotic dose of 1 gm Cefotaxime vial was administered followed by Dexamethasone phosphate (as sodium salt) 4 mg vial through peripheral IV route at the beginning of the procedure. A local anesthetic solution of Articaine 4% containing Epinephrine (1:200,000) was infiltrated along the proposed operative field for hemostasis.
* A three-line pyramidal incision was performed. The distal incision was carried buccally across the external oblique ridge, and then joined to a gingival incision running buccally around the necks of the teeth on which the guide rests. The releasing incision is carried in a curved manner inferiorly and anteriorly, keeping in mind not to extend to the area of the mental foramen. Reflection of the flap was done with a periosteal elevator beginning from under the periosteum of the anterior buccal incision, working parallel to the gingival margin to detach the papillae and push distally.
* Once the field of interest was exposed, the guide was introduced onto the bone and teeth, and moved until a tight fit was achieved throughout its fitting surface. When needed, the guide was secured to the underlying bones by 2.0 miniscrews placed through their preplanned guiding tubes.
* Via a small stab incision through the skin, a transbuccal trochar is introduced, through which the self-drilling extraoral distractor pins are passed. The pins are inserted into the mandible at their designated points of entry through the guide.
* Using a piezotome, the osteotomy line is marked and the osteotomy is initiated guided by the osteotomy slit in the guide. The fixating screws and the guide are then removed. The use of piezotome allowed the planning of the osteotomies through the path of the inferior alveolar nerve without fear of nerve injury.
* After guide removal, the osteotomy is completed. The distractor is connected to the extraoral distractor pins and is then activated to insure free mobility of the distal segment. Once confirmed, the distractor is returned to its zero position. The flap was then repositioned and closed using 4-0 Braided Polyglycolic Acid sutures.

ELIGIBILITY:
Inclusion Criteria:

1. Patients free from any disease affecting bone formation of both sexes was included in the study.
2. Patients younger than 25 years old.
3. Patients included in the study were hemifacial microsomia
4. Distraction range was between 15-20 mm.

Exclusion Criteria:

1. The presence of uncontrolled systemic disease.
2. Previous radiotherapy on head and neck region.
3. Chemotherapy within the past 12-month period.
4. An active infection at the distraction site.

Ages: 5 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2015-12-30 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Standard cephalometric parameters of cosmetic improvement will be assessed in Degree (0) unit | 6 months
  The surgery of distraction osteogenesis is unpredictable the aim of use of computer planning is to make the surgery predictable to improve cosmetic results. the results will be by fixed radio graphic parameters as SNA, ANB to evaluate improvement in mandibular position, mandibular plane angle and smile orientation for occlusal cant assessment, H-angle and position of H-line to assess the retrognathia of chin all measurment will be done in degree unit

CONTACTS AND LOCATIONS:
Overall Officials: yasser el hadidi, mds, Principal Investigator — Ain Shams University
Locations (1):
- Ain shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided